CLINICAL TRIAL: NCT02824796
Title: Group Training for Parents Whose Children Suffer From ADHD and Comorbidity Using a Behavioral-Dynamic Approach: A Randomized Controlled Trial
Brief Title: Group Training for Parents Whose Children Suffer From ADHD and Comorbidity Using a Behavioral-Dynamic Approach
Acronym: SPBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015096
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-01

CONDITIONS: ADHD
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schema Parent Behavioral Training (Experimental): An enhanced protocol which combines a Schema Focused Therapy (SFT) and Behavioral Parent Training (PBT)
  Interventions: Behavioral: Schema Parent Behavioral Training
- Parent Behavioral Training (Active Comparator): Usually medication & The usual PBT treatment
  Interventions: Behavioral: Parent Behavioral Training

INTERVENTIONS:
Behavioral: Schema Parent Behavioral Training — A novel protocol for parent whose children suffer from ADHD and comorbidities. The protocol combines elements from Schema Focus Therapy (SFT) and Parent Behavioral Training (PBT)
  Arms: Schema Parent Behavioral Training
Behavioral: Parent Behavioral Training — A state of the art Parent Behavioral Treatment (PBT) for Children who suffer from ADHD symptoms
  Arms: Parent Behavioral Training

SUMMARY:
The purpose of this study is to determine whether a new parent training protocol for children with Attention Deficit Hyperactivity Disorder (ADHD) can over perform the state of the art Parent Training protocol (PBT) by increasing the long term effectiveness of the treatment, reducing the dropout rate and reducing the comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Parents to children 6-12 with ADHD symptoms according to the criteria of Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-V)
* The child was diagnosed in the past as ADHD by MD

Exclusion Criteria:

* Parents with psychotic symptoms or suicidality
* Parents with active manic episode
* Parents with substance dependence
* Parents with autism spectrum disorder

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent-teacher-rated ADHD symptoms | baseline, 12 weeks, 25 weeks, 3 months, 6 months, 12 months
  The Child Behavior Checklist (CBCL)-Attention Problem Scale (Child Behavior Checklist)

SECONDARY OUTCOMES:
Dropout rate | baseline, 12 weeks, 25 weeks
  Group dropout rate during treatment
Change from baseline in parent-teacher-rated Comorbidities symptoms | baseline, 25 weeks, 3 months, 6 months, 12 months
  CBCL Internalizing score (Child Behavior Checklist)

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Children and Adolescent Clinic, Maccabi Health Services, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee PC, Niew WI, Yang HJ, Chen VC, Lin KC. A meta-analysis of behavioral parent training for children with attention deficit hyperactivity disorder. Res Dev Disabil. 2012 Nov-Dec;33(6):2040-9. doi: 10.1016/j.ridd.2012.05.011. Epub 2012 Jun 29. PMID 22750360
- [Derived] Solan M, Brunstein Klomek A, Ankori G, Bloch A, Apter A, Plishty S. Impact of a New Parent Behavioral-Schema Training on Children with ADHD: A Pragmatic Control Trial. J Atten Disord. 2021 Dec;25(14):2048-2059. doi: 10.1177/1087054720959711. Epub 2020 Sep 30. PMID 32996352